CLINICAL TRIAL: NCT05106907
Title: An Open and Single Dose-escalation Study to Evaluate the Safety and Clinical Activity of Allogeneic CAR-T Targeting CD19(ThisCART19) in Patients With Relapsed and/or Refractory Non-Hodgkin's B Cell Lymphoma (r/r B-NHL)
Brief Title: Safety and Clinical Activity of ThisCART19 in Patients With r/r Non-Hodgkin's B Cell Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundamenta Therapeutics, Ltd. (Industry)
Collaborators: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FT400-002
Record Dates: First submitted 2021-10-25; First posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: B-cell Malignancy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ThisCART19 cells injections (Experimental): In this study, allogeneic anti-CD19 CAR T Cells(ThisCART19 cells) is used to treat patients with refractory or relapsed CD19 positive B cell malignancies.
  Interventions: Biological: ThisCART19 cells

INTERVENTIONS:
Biological: ThisCART19 cells — 0.2-60 x 10^6 CAR T cells per kg body weight

SUMMARY:
A single arm, open-label, dose-escalation study to evaluate the safety and clinical activity of ThisCART19 (Allogeneic CAR-T targeting CD19) in patients with relapsed and/or refractory non-Hodgkin's B cell lymphoma (r/r B-NHL).

DETAILED DESCRIPTION:
ThisCART19 cell is a non-gene-editing allogeneic CAR-T cell targeting CD19. This study is designed to evaluate the safety and clinical activity of ThisCART19 in patients with CD19 positive, relapsed and/or refractory non-Hodgkin's B cell lymphoma (r/r B-NHL).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years old, no gender and race limited;
2. Estimated life expectancy > 12 weeks deemed by investigator；
3. CD19 were positive by histopathology and/or cytology diagnosis；
4. Patients with relapsed and/or refractory non-Hodgkin's B cell lymphoma (r/r B-NHL)；
5. Relevant indicators for disease or assessment within 4 weeks after the last treatment;
6. Quality of Life Score (KPS) >50%；
7. Subject has adequate organ function at screening, cardiac ejection fraction ≥ 40%, no evidence of pericardial effusion as determined by an echocardiogram (ECHO); serum ALT/ AST <3 upper limit of normal (ULN); bilirubin<2.0 mg/dl; serum creatinine ≤1.6 mg/dl and/or BUN ≤ 1.5 mg/dl;
8. No remission or relapse after hematopoietic stem cell transplantation or autologous somatic immunotherapy;
9. Unsuitable conditions for stem cell transplantation;
10. Signed informed consent form (ICF).

Exclusion Criteria:

1. Women in pregnancy or lactation;
2. In active infection including hepatitis B, hepatitis C, HIV, or other fatal viral and bacterial infection；
3. The absolute count of nonprimary neutrophil < 0.75×10^9/L or platelet count < 50×10^9/L;
4. Abnormal vital signs and failure to cooperate with examination;
5. Patients with mental or psychological diseases who cannot cooperate with treatment and efficacy evaluation;
6. Highly allergic constitution or history of severe allergy;
7. Patients with systemic infection or severe local infection requiring anti-infection treatment;
8. Patients with severe autoimmune diseases;
9. Presence of any other conditions that are unsuitable for this study as judged by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-10-25 (Actual); Primary Completion 2023-10-24 (Estimated); Study Completion 2024-10-24 (Estimated)

PRIMARY OUTCOMES:
Treatment related adverse events | 90 days post infusion
  Incidence and severity of adverse events as assessed by NCI-CTCAE 5.0

SECONDARY OUTCOMES:
Overall Remission Rate (ORR) | up to 90 days
  Anti-tumor efficacy by 2014 Lugano criteria
Progression free survival time | 3 years
  The interval between administration and disease progression or death
Overall survival time | 3 years
  The interval between administration and death caused by any reason
Event-free survival (EFS) | 3 years
  EFS is calculated from administration to death, progression of the disease, relapse or gene recurrence, whichever comes first, or last visit.

CONTACTS AND LOCATIONS:
Overall Officials: Zhengyu Li, Ph.D, Study Chair — The Affiliated Hospital of Xuzhou Medical University
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China